CLINICAL TRIAL: NCT02394353
Title: Impact of Bariatric Surgery on the Evolution of Nonalcoholic Fatty Liver Disease: a Comparative Clinical Trial Between Sleeve Gastrectomy and Gastric Bypass
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, Fernando de Barros, Fernando de Barros, Ministry of Health, Brazil
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Interventions
Record Dates: First submitted 2015-03-04; First posted 2015-03-20 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Obesity; Fatty Liver
Keywords: bariatrics; transient elastography
MeSH Terms: conditions — Obesity; Fatty Liver

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sleeve Gastrectomy (Active Comparator): Patients undergoing the sleeve gastrectomy surgery
  Interventions: Device: Transient hepatic elastography
- Gastric Bypass (Active Comparator): Patients undergoing the gastric bypass surgery
  Interventions: Device: Transient hepatic elastography

INTERVENTIONS:
Device: Transient hepatic elastography

SUMMARY:
Aim: To compare prospectively two bariatric surgery techniques: sleeve gastrectomy (SG) vs gastric bypass (GB) in the evolution of nonalcoholic fatty liver disease (NAFLD) measured by the transient elastography in the first year. Methods: This is a randomized clinical trial with morbidly obese patients, between 18-60 years old from a Federal Hospital, Ministry of Health, Brazil. Patients were divided into 2 groups: group 1 - SG (n = 30) and group 2 - GB (n = 30). The randomization was made by lots. In the GB the investigators created 30 ml pouch, with a pancreatic and an alimentary limb of 1 meter, and a calibrated gastroenterostomy (1.5 cm diameter). In SG the investigators calibrated the gastric tube with a bougie number 32 (70 ml). The variables were compared one week before surgery and in the postoperative time (1, 3, 6 and 12 months). The variables were: patient anthropometry, laboratory tests and the transient liver elastography.

ELIGIBILITY:
Inclusion Criteria:

The eligibility criteria was:

* morbid obesity patient grade II or grade III (BMI > 35) in prepare to bariatric surgery.

Exclusion Criteria:

The exclusion criteria were:

* age under 18 years or greater than 65 years old,
* chronic diseases (heart failure, chronic liver disease), and
* alcohol abuse (abuse was considered in those who consume more than 14 drinks per week).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Measure of fatty liver disease by transient hepatic elastography | Participants will be followed an average of 3 months
  Tha aim is to compare the evolution of the fatty liver disease between the sleeve gastrectomy and gastric bypass

SECONDARY OUTCOMES:
Transversal study comparing comorbidities and transient hepatic elastography | Participants will be submitted a correlation with comorbidities
  Tha aim is to find some relationship

OTHER OUTCOMES:
Prevalence of advanced fibrosis in assyntomatic obese patients | Fibrosis will be assessed by transient hepatic elastography in the pre-operative period
  Tha aim is identified patients with advanced disease

CONTACTS AND LOCATIONS:
Locations (1):
- Fluminense Federal University, Niterói, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] de Barros F, Setubal S, Martinho JM, Leite NC, Guarana T, Monteiro ABS, Villela-Nogueira CA. The Correlation Between Obesity-Related Diseases and Non-alcoholic Fatty Liver Disease in Women in the Pre-operative Evaluation for Bariatric Surgery Assessed by Transient Hepatic Elastography. Obes Surg. 2016 Sep;26(9):2089-2097. doi: 10.1007/s11695-016-2054-y. PMID 26803754
- [Derived] de Barros F, Setubal S, Martinho JM, Monteiro AB. Early Endocrine and Metabolic Changes After Bariatric Surgery in Grade III Morbidly Obese Patients: A Randomized Clinical Trial Comparing Sleeve Gastrectomy and Gastric Bypass. Metab Syndr Relat Disord. 2015 Aug;13(6):264-71. doi: 10.1089/met.2014.0152. Epub 2015 Apr 28. PMID 25919069